CLINICAL TRIAL: NCT06738563
Title: Impact of Breast Milk on the Infectivity and Transmission of Different Viruses "BREASTMILKVIR"
Acronym: BREASTMILKVIR
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-017; 2024-A01159-38 (Other: ID-RCB)
Record Dates: First submitted 2024-12-04; First posted 2024-12-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-12

CONDITIONS: Breastmilk Collection
Keywords: Milk; Maternal; Virus; Transmission; Infectivity
MeSH Terms: conditions — Breast Milk Expression; Virus Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactating women: Lactating adult women who donate their milk
  Interventions: Other: Collection breast milk

INTERVENTIONS:
Other: Collection breast milk — Collection of a milk sample taken as part of women's donation

SUMMARY:
Exclusive breastfeeding during the first six months of life and continued breastfeeding for at least 24 months constitute the optimal feeding method for infants and young children.

However, breast milk and breastfeeding can be significant pathways for the transmission of certain viruses.

The objective of this study is to examine the influence of human breast milk and its composition on viral infectivity and viral transmission of the HTLV-1 virus and arboviruses such as Zika virus, yellow fever, dengue, and tick-borne encephalitis.

DETAILED DESCRIPTION:
Exclusive breastfeeding during the first six months of life and continued breastfeeding for at least 24 months constitute the optimal feeding method for infants and young children.

However, breast milk and breastfeeding can be significant pathways for the transmission of at least three human viruses: HTLV-1, HIV, and human cytomegalovirus (CMV).

To address the following main objective: to study the influence of human breast milk and its composition on viral infectivity and viral transmission of the HTLV-1 virus and arboviruses such as Zika virus, yellow fever, dengue, and tick-borne encephalitis.The study plans to collect milk samples from lactating women who are registered with the Lactarium of Île-de-France to donate their breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Female gender
* Lactarium Ile-de-France donors
* Subjects covered by a Social Security scheme, excluding State Medical Aid

No inclusion criteria:

- Women opposing participation in the study

Exclusion Criteria:

- Positive HIV, HBV, HCV and HTLV serologies (Lactarium exclusion criteria)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Breastfeeding adult women who register with the Île-de-France Milk Bank to donate their milk.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Study the influence of breast milk and its composition on viral infectivity and oral transmission of HTLV-1 and arboviruses such as Zika virus, yellow fever virus, dengue virus, and tick-borne encephalitis virus. | 36 months
  Various viruses will be incubated with milk samples. The influence of milk on the different viruses will be studied. The capacity of these viruses incubated with milk to infect the target cells (immune or epithelial cells, depending on the virus) will be measured (measurement of the number of infected cells).

SECONDARY OUTCOMES:
Determine the antiviral or proviral mechanisms of certain biological factors in breast milk. | 36 months
  The level of proteins, carbohydrates and fatty acids will be measured in the milk using an infrared spectrometer. The aim is to find out whether the composition of the milk can influence its antiviral or proviral mechanisms.
Determine the role of breast milk in the mechanisms by which the relevant viruses cross an epithelium. | 36 months
  Following the addition of viral particles or infected cells to the apical side of an "in vitro" intestinal model, the impact of breastmilk on crossing efficacy and underlying mechanisms will be assessed.
  Measurement of the number of viruses that cross the barrier of the intestinal epithelium in the presence of milk by comparing the number of viruses that cross the barrier of the intestinal epithelium without being incubated with milk.
Determine the influence of a few hours of incubation at 4°C (refrigeration) on the previously mentioned mechanisms. | 36 months
  Milk samples will be incubated at 4°C. It has been demonstrated for several enveloped viruses, including the Zika virus, that refrigeration of breast milk (4°C) induces an antiviral effect. However, some experiments seem to indicate major differences in the kinetics of this effect, depending on milk factors. Kinetics will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie RIGOURD, Dr, Principal Investigator — Lactarium Ile-de-France, Necker-Enfents Malades Hospital
Locations (1):
- Lactarium Ile-de-France, Necker-Enfents Malades Hospital, Paris, France